CLINICAL TRIAL: NCT03724877
Title: Comparative Effectiveness of Triple Therapy in COPD: A New-user Cohort Study
Brief Title: Effectiveness of Triple Therapy in COPD
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1237-0078
Record Dates: First submitted 2018-10-29; First posted 2018-10-30 (Actual); Results first posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects with Chronic obstructive pulmonary disease (COPD)
  Interventions: Drug: Long-acting beta2-agonist-long-acting muscarinic antagonists-inhaled corticosteroids(LABA-LAMA-ICS); Drug: Long-acting beta2-agonist-inhaled corticosteroids-long-acting muscarinic antagonists (LABA-LAMA)

INTERVENTIONS:
Drug: Long-acting beta2-agonist-long-acting muscarinic antagonists-inhaled corticosteroids(LABA-LAMA-ICS) — (LABA-LAMA-ICS)
Drug: Long-acting beta2-agonist-inhaled corticosteroids-long-acting muscarinic antagonists (LABA-LAMA) — (LABA-LAMA)

SUMMARY:
To assess the effectiveness of maintenance treatment of Chronic obstructive pulmonary disease (COPD) with the Long-acting beta2-agonist - long-acting muscarinic antagonists-inhaled corticosteroids (LABA-LAMA-ICS) combination with a LABA-LAMA combination on the risk of COPD exacerbation and the safety on the incidence of community acquired pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* New users of long-acting bronchodilators, Long-acting beta2-agonist (LABA) and long-acting muscarinic antagonists (LAMA) on the same date or of LABA, LAMA and inhaled corticosteroids (ICS), either as a fixed-dose combination (LABA-ICS) or free combination, on the same date between January 2002 and December 2016.
* Diagnosis of Chronic obstructive pulmonary disease (COPD) prior to first maintenance inhaler and age ≥ 55 years at first maintenance inhaler.

Exclusion Criteria:

* Less than one year of medical history information prior to the date of combined treatment initiation (study cohort entry)
* Asthma diagnosis prior to study cohort entry

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Incident new-user cohort design with high-dimensional propensity scores to match the two comparison groups of COPD.
Sampling Method: Non-Probability Sample
Enrollment: 8853 (Actual)
Dates: Start 2018-11-10 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2018-11-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Practice Research Datalink, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions: 1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). Requestors can use the following link http://trials.boehringer-ingelheim.com/ to:
  1. find information in order to request access to clinical study data, for listed studies.
  2. request access to clinical study documents that meet criteria, and upon a signed 'Document Sharing Agreement.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Base cohort consisted participants with ChronicObstructivePulmonaryDisease(COPD) who subsequently received at least one prescription for a long-acting bronchodilator, either Long-Acting Beta2-Agonist(LABA) or long-acting MuscarinicAntagonists(LAMA), or for inhaled corticosteroid(ICS), alone or in combination, from 1January2002 until 31December2015.
Pre-assignment Details: Population-based incident new-user cohort design with high-dimensional time-conditional propensity score matching. The study cohort was formed from the base cohort using an incident new-user cohort design with time-conditional propensity scores.
Groups:
- LABA-LAMA-ICS: The participants with COPD initiating treatment with LABA-LAMA-ICS combination as three or two inhalers on the same day were included in this group. Participants were followed for up to one year from the cohort entry date, the date of death, 31 March 2016, or the end of coverage in the practice, whichever occurred first.
- LABA-LAMA: The participants with COPD with their first concurrent prescriptions of a LAMA and LABA (no ICS) as two inhalers on the same day included in this group were matched on high-dimensional propensity score with patients initiating treatment with LABA-LAMA-ICS combination as three or two inhalers on the same day. Participants were followed for up to one year from the cohort entry date, the date of death, 31 March 2016, or the end of coverage in the practice, whichever occurred first.
Period: Overall Study
Arm/Group | LABA-LAMA-ICS | LABA-LAMA
Started (Started are Initiators) | 6921 | 1932
Completed | 6921 | 1932
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The main analysis was on matched patients. The cohort of initiators of LAMA-LABA-ICS and their propensity score-matched initiators of LAMA-LABA.
Groups:
- Total: Total of all reporting groups
Arm/Group | LABA-LAMA-ICS | LABA-LAMA | Total
Number analyzed (Participants) | 6921 | 1932 | 8853
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.9 (8.5) | 71.6 (8.5) | 71.8 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2619 | 746 | 3365
  Male | 4302 | 1186 | 5488
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Hospitalised With Severe Exacerbation
Description: The primary outcome event for effectiveness was the first COPD exacerbation to occur after cohort entry. The event was defined as a hospitalization with a primary diagnosis of COPD (severe exacerbation) is presented.
Time Frame: 1 year
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | LABA-LAMA-ICS | LABA-LAMA
Number analyzed (Participants) | 6921 | 1932
Participants | 3074 | 630
Statistical Analysis 1: Comparison: LABA-LAMA-ICS vs LABA-LAMA; Test type: Other; Regression, Cox; Adjusted hazard ratio (HR) = 1.04, 95% CI 2-sided [0.79 to 1.38] — After matching on high-dimensional propensity scores, sex prior severe exacerbation, prior maintenance treatment and calendar time, adjusted further for the deciles of propensity score and percent predicted forced expiratory volume1 (FEV1)

2. Primary Outcome: Number of Participants Hospitalised With Moderate Exacerbation
Description: The primary outcome event for effectiveness was the first COPD exacerbation to occur after cohort entry. The event was defined as a hospitalization with the prescription of an oral corticosteroid, namely prednisolone (moderate exacerbation) is presented.
Time Frame: 1 year
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | LABA-LAMA-ICS | LABA-LAMA
Number analyzed (Participants) | 6921 | 1932
Participants | 2487 | 542
Statistical Analysis 1: Comparison: LABA-LAMA-ICS vs LABA-LAMA; Test type: Other; Regression, Cox; Adjusted HR = 0.97, 95% CI 2-sided [0.87 to 1.09] — After matching on high-dimensional propensity scores, sex prior severe exacerbation, prior maintenance treatment and calendar time, adjusted further for the deciles of propensity score and percent predicted FEV1

3. Primary Outcome: Number of Participants Hospitalised With Community-acquired Pneumonia (Serious Pneumonia)
Description: The primary outcome event for safety was the occurrence of the first hospitalization for community-acquired pneumonia (serious pneumonia).
Time Frame: 1 year
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | LABA-LAMA-ICS | LABA-LAMA
Number analyzed (Participants) | 6921 | 1932
Participants | 3099 | 634
Statistical Analysis 1: Comparison: LABA-LAMA-ICS vs LABA-LAMA; Test type: Other; Regression, Cox; Adjusted HR = 1.46, 95% CI 2-sided [1.03 to 2.07] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: The Rate of COPD Exacerbations Over the One-year Follow-up
Description: This outcome was based on the number of hospitalizations and on the number of courses of treatment with an oral corticosteroid. A gap of at least 30 days between treatment courses was required to consider the exacerbations as separate events.
Time Frame: 1 year
Population: as for baseline characteristics
Measure: Number; unit: exacerbations per 100 person year
Arm/Group | LABA-LAMA-ICS | LABA-LAMA
Number analyzed (Participants) | 6921 | 1932
exacerbations per 100 person year
  Moderate/ sever exacerbation | 94.4 | 89.3
  Severe exacerbation | 13.4 | 11.0
Statistical Analysis 1: Comparison: LABA-LAMA-ICS vs LABA-LAMA; Moderate/ sever exacerbation; Test type: Other; Negative binomial regression model; Adjusted rate ratio = 0.93, 95% CI 2-sided [0.83 to 1.04] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: LABA-LAMA-ICS vs LABA-LAMA; Severe exacerbation; Test type: Other; Negative binomial regression model; Adjusted rate ratio = 0.94, 95% CI 2-sided [0.70 to 1.28] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event information was not applicable for this study.
Description: This was an observational study and was not designed to assess adverse event; therefore safety reporting was not applicable for this study. Adverse Events were not monitored/assessed.
Arm/Group | LABA-LAMA-ICS | LABA-LAMA
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/77/NCT03724877/Prot_SAP_000.pdf